CLINICAL TRIAL: NCT01886703
Title: Feasibility of a Supported Walking Program for Breast and Head-and-Neck Cancer Survivors Receiving Adjuvant Radiation Therapy
Brief Title: Feasibility of a Walking Program for Cancer Survivors Receiving Radiation Therapy
Acronym: PEDWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Margie McNeely, Assistant Professor, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ACREC 26059
Record Dates: First submitted 2013-06-16; First posted 2013-06-26 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Physical Activity
Keywords: Physical activity; Exercise; Quality of Life; Radiation Therapy; Breast Cancer; Head and Neck Cancer
MeSH Terms: conditions — Motor Activity; Breast Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Walking Intervention (Experimental): Pedometer Walking Program
  Interventions: Behavioral: Pedometer Walking Program

INTERVENTIONS:
Behavioral: Pedometer Walking Program — All subjects will be prescribed a low-intensity walking program based on their current activity level and an daily assigned step count goal (with the current physical activity recommendations of 30 minutes of moderate-to-vigorous activity per day or 150 minutes per week as the ideal goal). Participants will be provided with face-to-face counseling and written material describing their specific individualized walking program. Participants will also be instructed to maintain their normal activities as much as possible during the intervention period. Participants will be given a pedometer and instructed to wear it at least 5 days per week for the duration of the study.

SUMMARY:
This pilot study will assess whether a supported pedometer-based walking program is helpful in maintaining physical activity for breast and head-and-neck cancer patients who are undergoing radiation therapy. Follow-up monitoring sessions will be scheduled to help provide support for physical activity during radiation therapy. We will also examine the relationship of physical activity and quality of life outcomes to help inform future research.

DETAILED DESCRIPTION:
Will the integration of a patient-centered exercise prescription and supportive counseling attenuate declines in physical activity during radiation therapy? To address this question, this study will assess the feasibility of a patient-centered walking program for breast and head-and-neck cancer patients undergoing radiation therapy. Follow-up monitoring sessions will be scheduled to help provide support and ongoing counseling to facilitate increased activity (through walking) during radiation therapy. We will also examine the effect of the walking program on other outcomes such as happiness, depression and sleep to determine point estimates and measures of variability to inform future research.

ELIGIBILITY:
Inclusion Criteria:

* Survivors with a diagnosis of breast cancer or head and neck cancer
* Adults aged 18 years or older
* Commencing adjuvant radiation therapy treatments
* Karnofsky Performance Status greater than or equal to 60%

Exclusion Criteria:

* Clinical or radiological evidence of active disease, either local or metastatic
* Serious non-malignant disease, such as cardiac failure or advanced arthritis of weight bearing joints, which would preclude daily treatment and follow-up
* Patients for whom physical activity or exercise is contraindicated
* Psychiatric or addictive disorders which preclude obtaining informed consent or adherence to the protocol
* Unable to comply with the protocol, measurement and follow-up schedule (e.g., scheduling conflicts, time commitment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Accrual Rate and Completion Rate | Anticipated duration of radiation therapy of 6 weeks
  Accrual: Number of participants agreeing to participate divided by the number of eligible participants Completion rate: number of participants completing the trial

SECONDARY OUTCOMES:
Adherence | Anticipated duration of radiation therapy of 6 weeks
  Adherence to the intervention protocol: number of days meeting target step count

OTHER OUTCOMES:
6-Minute Walk Test | Change from baseline to anticipated end of radiation therapy of 6 weeks
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a six minutes time period on a hard, flat surface (e.g., 100 foot hallway).
Physical Activity | Change from baseline to anticipated duration of radiation therapy of 6 weeks
  An accelerometer armband will be used to provide a breakdown of an individual's daily activity.
Self-esteem | Change from baseline to anticipated duration of radiation therapy of 6 weeks
  Rosenberg Self-Esteem Scale (10 item)
Depression | Change from baseline to anticipated duration of radiation therapy of 6 weeks
  Beck Depression Inventory II (21 item)
Happiness | Change from baseline to anticipated duration of radiation therapy of 6 weeks
  Oxford Happiness Questionnaire (29 items)
Sleep | Change from baseline to anticipated duration of radiation therapy of 6 weeks
  Pittsburgh Sleep Quality Index (9 item)
Fatigue | Recorded daily during study period of 6 weeks
  Visual analogue scale, recorded as part of daily diary

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNeely, PhD, Principal Investigator — University of Alberta and Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
No plan in place